CLINICAL TRIAL: NCT04637958
Title: Correlation Between Femoral Head and Cup Size and Postoperative Pain in Total Hip Arthroplasty
Acronym: jantje
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Research Orthopedie, Research, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: JBFemHeadTHP; UZ Leuven (Other: UZ Leuven)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Femoral Head Size; Cup Size THP; Postoperatie Groin Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pain: THA
  Interventions: Device: THA
- no pain: THA
  Interventions: Device: THA

INTERVENTIONS:
Device: THA — Total hip arthroplasty

SUMMARY:
We want to investigate the correlation between the native femoral head and the implanted cup in Total hip arthroplasty. As second parameter to investigate we believe an oversized cup will cause groin pain. We want to find a cutoff value to predict groin pain after cup implementation in THA.

ELIGIBILITY:
Inclusion Criteria:

* all primary THA

Exclusion Criteria:

* DDH-LCP
* Acetabulum/femoral neck fracture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: retrospective database THA
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Correlation between femoral head and cup size and postoperative pain in Total Hip arthroplasty | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Background] Odri GA, Padiolleau GB, Gouin FT. Oversized cups as a major risk factor of postoperative pain after total hip arthroplasty. J Arthroplasty. 2014 Apr;29(4):753-6. doi: 10.1016/j.arth.2013.07.001. Epub 2013 Aug 6. PMID 23927907